CLINICAL TRIAL: NCT03213366
Title: Empowering With PrEP Cluster-Randomized Controlled Trial: A Social Media Based Peer-Led Intervention for HIV Prevention
Brief Title: Social Media Based Peer-Led Intervention for HIV Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Albert Einstein College of Medicine (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Viraj V. Patel, Assistant Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016-7263; 5K23MH102118-04 (NIH)
Record Dates: First submitted 2017-03-28; First posted 2017-07-11 (Actual); Results first posted 2019-09-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: HIV Prevention; PrEP Uptake
Keywords: PrEP; HIV prevention; Public Health Social Media Campaign; Peer Intervention

STUDY DESIGN:
Intervention Model Description: There will be two groups of Peer Leaders recruited. One group of Peer Leaders will be randomized to deliver the E-PrEP intervention and the second group of peer leaders will be randomized to deliver a general health campaign (control).
Who Masked: Participant, Outcomes Assessor
Masking Description: Both Peer Leaders and participants will be masked to the group randomized to. The statistician, who will be analyzing the data, will also be masked to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-PrEP- Peer-Led Intervention about PrEP (Experimental): 8 Peer Leaders (PLs) will be randomly assigned to the E-PrEP arm. Each of the PLs will recruit at least 15 participants into a private social media group on one of several social media platforms. PLs will then deliver a behavioral intervention over a 6 week period, posting information and engaging participants in a discussion about PrEP, PrEP access, and other related health issues. All contents will be formatted to be both mobile device accessible.
  Interventions: Behavioral: E-PrEP- Peer-Led Intervention about PrEP
- BxNow - General Health Campaign (Active Comparator): BxNow is an attention-matched control. Eight of the 16 PLs will be randomly assigned to the BxNow arm. The BxNow campaign will be a 6-week long social media intervention about general health wellness topics chosen and administered by the PLs assigned into this arm. Similarly to the intervention group, PLs in the BxNow arm will create private social media groups and recruit participants into these private groups. General health information in the BxNow arm will be posted with the same frequency as in the intervention arm.
  Interventions: Behavioral: BxNow - General Health Campaign

INTERVENTIONS:
Behavioral: E-PrEP- Peer-Led Intervention about PrEP — Intervention contents and targets were informed by a systematic review of PrEP barriers and facilitators, a locally conducted qualitative study, and key informant and peer leader inputs. The contents were developed or adapted by study staff and peer leaders. Components and associated text have been designed to engage participants in online discussions about PrEP and related health and social topics. Posts will also include information about linkage-to-care, and insurance access. New contents will be posted almost daily.
  Arms: E-PrEP- Peer-Led Intervention about PrEP
Behavioral: BxNow - General Health Campaign — BxNow will focus on general health topics unrelated to HIV or sexual health (i.e. fitness, nutrition, smoking), as chosen by PLs. Contents will be developed or adapted by PLs and posted almost daily. Posts will also include information about linkage-to-care and insurance access. At the end of the intervention, BxNow participants will be exposed to E-PrEP components at the end of the trial.
  Arms: BxNow - General Health Campaign

SUMMARY:
The purpose of this study is to test the feasibility, acceptability, and preliminary efficacy of E-PrEP on reaching young men of color who have sex with men (YMCSM) at high-risk of HIV infection to reduce HIV acquisition. E-PrEP is a peer-designed social media-based health intervention to increase PrEP awareness, knowledge, and motivation as a tool for HIV prevention and to increase linkage to primary care.

DETAILED DESCRIPTION:
This study examines a social media based peer-led and delivered intervention focused on increasing PrEP adoption in young men of color who have sex with men (YMCSM). While prior efficacy trials have included YMCSM 18-29, we will focus on PrEP in YMCSM outside clinical trial settings. Rather than an alternative medium for implementation of existing interventions designed for in-person contact, social media may be a true 'game changer' to engage hard to reach individuals. While many online behavioral interventions exist, including some that use social media, this will be one of the few studies to use and test social media to facilitate uptake of a biomedical intervention. E-PrEP will connect the target population (YMCSM) to a new prevention tool (PrEP) through rapid linkage to medical care, accelerating diffusion of PrEP. Given the paucity of data regarding social media-based interventions to change health-related behavior, E-PrEP may have a marked impact on future bio-behavioral interventions, especially those that include diffusion of innovation. Social media offers the power of scale and efficiency for large potential impact, even with relatively low-intensity interventions. Similarly, PrEP, if widely adopted in high-risk populations and offered with behavioral interventions, could markedly decrease HIV infection rates. Social media-based, peer-led approaches like E-PrEP could be used to enhance efforts by community-based and other organizations that employ internet-assisted or peer-outreach strategies to improve health.

Primary Aim: To test the feasibility and preliminary efficacy of E-PrEP for increasing PrEP adoption in a cluster-randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or Transgender individual; Ages 18-29; Have had unprotected anal sex with a male partner in the prior 12 months; Fluent in English or Spanish; Are HIV-negative or unknown status (self-report); Identify as Black and/or Latino

Exclusion Criteria:

* YMCSM who do not consent/assent to study; not currently using at least one of 2 social media sites that will be used for the E-PrEP intervention (not using Facebook, or Instagram), and do not live in New York City.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Including participants who self-identify as male or transgender individual and also have sex with men.
Enrollment: 152 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viraj Patel, MD, MPH, Principal Investigator — Montefiore Medical Center
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel VV, Ginsburg Z, Golub SA, Horvath KJ, Rios N, Mayer KH, Kim RS, Arnsten JH. Empowering With PrEP (E-PrEP), a Peer-Led Social Media-Based Intervention to Facilitate HIV Preexposure Prophylaxis Adoption Among Young Black and Latinx Gay and Bisexual Men: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2018 Aug 28;7(8):e11375. doi: 10.2196/11375. PMID 30154071

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Peers
Groups:
- E-PrEP- Peer-Led Intervention About PrEP: We recruited Peer Leaders over a 5-week period and then randomly assigned them to the 2 arms. Peer Leaders were blinded to their study condition. Peer leaders recruited study participants via their existing online social networks to complete an online eligibility screener and baseline survey. Study participants were then directed to join a private online group, facilitated and moderated by the peer leader who had recruited them.
  Content: The E-PrEP campaign focused on delivering information about PrEP. The materials were composed of 6 weeks of publicly available PrEP educations materials selected by peer advisors prior to the intervention (i.e. information on how to talk to your doctor about PrEP, where to get PrEP, side effects, etc.). The materials mapped out onto Diffusion of Innovation (DOI) and Information, Motivation, Behavior (IMB) domains. Peer leaders framed the E-PrEP materials in their own words when posting the materials to their online private group.
- BxNow-General Health Control Arm:: We recruited Peer Leaders over a 5-week period and then randomly assigned them to the 2 arms. Peer Leaders were blinded to their study condition. Peer leaders recruited study participants via their existing online social networks to complete an online eligibility screener and baseline survey. Study participants were then directed to join a private online group, facilitated and moderated by the peer leader who had recruited them.
  Content: BxNow focused on a broad range of health topics prioritized by the peer leaders assigned to this arm, but did not include any contents about HIV or PrEP (i.e. depression, anxiety, suicide, intimate partner violence, drug use, awareness of sexually transmitted infections). BxNow was attention matched to the E-PrEP intervention timeline (6 weeks of materials) for both time and day of posts and frequency of posts. As with E-PrEP, standardized BxNow contents were delivered by peer leaders, framed using their own words.
Period: Overall Study
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow-General Health Control Arm:
Started | 81; 7 Peers | 71; 5 Peers
Completed | 72; 5 Peers | 67; 5 Peers
Not Completed | 9; 2 Peers | 4; 0 Peers
Not completed — Lost to Follow-up | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- BxNow- General Health Control Arm: We recruited Peer Leaders over a 5-week period and then randomly assigned them to the 2 arms. Peer Leaders were blinded to their study condition. Peer leaders recruited study participants via their existing online social networks to complete an online eligibility screener and baseline survey. Study participants were then directed to join a private online group, facilitated and moderated by the peer leader who had recruited them.
  Content: BxNow focused on a broad range of health topics prioritized by the peer leaders assigned to this arm, but did not include any contents about HIV or PrEP (i.e. depression, anxiety, suicide, intimate partner violence, drug use, awareness of sexually transmitted infections). BxNow was attention matched to the E-PrEP intervention timeline (6 weeks of materials) for both time and day of posts and frequency of posts. As with E-PrEP, standardized BxNow contents were delivered by peer leaders, framed using their own words.
- Total: Total of all reporting groups
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow- General Health Control Arm | Total
Number analyzed (Participants) | 81 | 71 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.28 (2.83) | 23.32 (3.39) | 23.84 (2.83)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identity: Male | 68 | 64 | 132
  Gender Identity: Female/Transfemale | 7 | 3 | 10
  Gender Identity: Transmale | 1 | 0 | 1
  Gender Identity: Gender Non-conforming/Gender Non-Binary | 2 | 0 | 2
  Gender Identity: Queer | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Latinx/Hispanic | 26 | 47 | 73
  Race/Ethnicity: Non-Hispanic Black | 55 | 24 | 79
Residence [Count of Participants; unit: Participants]
  Bronx | 44 | 35 | 79
  Brooklyn | 18 | 14 | 32
  Manhattan | 16 | 13 | 29
  Queens | 2 | 8 | 10
  Staten Island | 1 | 1 | 2
Sexual Identity [Count of Participants; unit: Participants]
  Gay/Homosexual | 60 | 56 | 116
  Queer | 12 | 3 | 15
  Bisexual | 7 | 10 | 17
  Heterosexual/Straight | 1 | 1 | 2
  Other | 1 | 1 | 2
Education Level [Count of Participants; unit: Participants]
  High School or Less | 36 | 27 | 63
  Some College | 28 | 35 | 63
  College and Beyond | 17 | 9 | 26
Employment [Count of Participants; unit: Participants] — Participants had the option to select more than one answer in order to best describe their employment status (not mutually exclusive).
  Participants
    Full Time | 24 | 29 | 53
    Part Time | 17 | 15 | 32
    Unemployed | 31 | 15 | 46
    Disable | 3 | 2 | 5
    Student | 12 | 13 | 25
Income [Count of Participants; unit: Participants]
  None | 12 | 14 | 26
  Less than $10,000 | 26 | 15 | 41
  $10,000-$19,999 | 11 | 10 | 21
  $20,000-$29,999 | 13 | 6 | 19
  $30,000-$39,999 | 11 | 16 | 27
  $40,000-more | 8 | 10 | 18
Living Situation [Count of Participants; unit: Participants]
  Don't have a place to live | 4 | 2 | 6
  Temporary Living Situation | 15 | 7 | 22
  Parents/Family | 29 | 36 | 65
  Partner/Boyfriend/Husband | 2 | 7 | 9
  Roomates | 20 | 14 | 34
  Alone | 11 | 4 | 15
  Wife/Females Partner/Girlfriend | 0 | 1 | 1
Health Insurance [Count of Participants; unit: Participants]
  Yes | 61 | 59 | 120
  No | 18 | 10 | 28
  I don't kno | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Intending to Start Using PrEP Over Time
Description: This primary outcome is intention to use PrEP in the next month measured at baseline, 6 weeks, and 12 weeks. This was assessed with a yes/no question (dichotomous variable). However, this variable does not include anyone who reported PrEP use at either 6 or 12 weeks.
  This outcome will inform sample size calculations for a subsequent fully powered trial.
Time Frame: baseline, 6 weeks, and 12 weeks
Population: Each of the rows indicates the number of participants who indicated intending to use PrEP at each time point (Baseline vs. 6 weeks vs. 12 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow- General Health Control Arm
Number analyzed (Participants) | 65 | 63
Participants
  Baseline: Yes | 32 | 34
  Baseline: No | 33 | 29
  6 Weeks: Yes | 23 | 27
  6 Weeks: No | 42 | 36
  12 Weeks: Yes | 27 | 32
  12 Weeks: No | 38 | 31
Statistical Analysis 1: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 6 weeks; Test type: Superiority; p = 0.5783, Mixed Models Analysis; Slope = -0.0095, 95% CI 2-sided [-0.04676 to 0.02776]
Statistical Analysis 2: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 12 weeks; Test type: Superiority; p = 0.3185, Mixed Models Analysis; Slope = -0.01692, 95% CI 2-sided [-0.05318 to 0.01933]

2. Primary Outcome: Number of Participants Using PrEP Over Time
Description: This outcome is the number of participants who self-report using PrEP at baseline, 6 weeks, or 12 weeks. This was measure by a yes/no question asking if the participant currently uses PrEP (dichotomous variable).
Time Frame: at baseline, 6 weeks, and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow- General Health Control Arm
Number analyzed (Participants) | 65 | 63
Participants
  Baseline: Yes | 13 | 11
  Baseline: No | 52 | 52
  6 weeks: Yes | 17 | 11
  6 weeks: No | 48 | 52
  12 weeks: Yes | 14 | 13
  12 weeks: No | 51 | 50
Statistical Analysis 1: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 6 weeks; Test type: Superiority; p = 0.07863, Mixed Models Analysis; Slope = 0.03674, 95% CI 2-sided [-0.00516 to 0.07863]
Statistical Analysis 2: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 12 weeks; Test type: Superiority; p = 0.1999, Mixed Models Analysis; Slope = 0.02594, 95% CI 2-sided [-0.01648 to 0.06836]

3. Secondary Outcome: Change in PrEP Knowledge
Description: Self-reported PrEP related knowledge.
  Participants were asked two questions about PrEP knowledge. For each question, they got one point if the answer was correct.
  Scale range from 0-2. The score were added and the average of the sum was reported.
  The higher the score, the higher the knowledge of PrEP.
Time Frame: at baseline, 6 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow- General Health Control Arm
Number analyzed (Participants) | 65 | 63
score on a scale
  Baseline | 1.86 (0.43) | 1.7 (0.59)
  6 Weeks | 1.86 (0.39) | 1.83 (0.46)
  12 Weeks | 1.83 (0.49) | 1.73 (0.55)
Statistical Analysis 1: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 6 weeks; Test type: Superiority; p = 0.8963, Mixed Models Analysis; Slope = 0.000443
Statistical Analysis 2: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 12 weeks; Test type: Superiority; p = 0.3229, Mixed Models Analysis; Slope = 0.004308

4. Secondary Outcome: PrEP Awareness
Description: Awareness about PrEP.
  PrEP awareness was measured with one question, scored 1 to 5. The mean for each arm was calculated at each time point.
  The higher the score, the higher the level of awareness about PrEP.
Time Frame: baseline, 6 weeks, 12 weeks
Population: T
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow- General Health Control Arm
Number analyzed (Participants) | 65 | 63
score on a scale
  Baseline | 4.14 (0.95) | 4.02 (0.88)
  6 Weeks | 4.29 (0.96) | 4.13 (0.91)
  12 Weeks | 4.52 (0.69) | 4.19 (0.91)
Statistical Analysis 1: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; Test type: Superiority; p = 0.2433, Mixed Models Analysis — This t-test was for the random effects model not for comparing the difference between the arms; Slope = 0.008705
Statistical Analysis 2: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 12 weeks; Test type: Superiority; p = 0.0839, Mixed Models Analysis; Slope = 0.01358

5. Secondary Outcome: PrEP Stigma
Description: Any stigma the participant might have about PrEP or those who use PrEP
  To measure PrEP Stigma we asked 3 questions, using a Likert scale (from 1-4; 1= Strongly Disagree, 4=Strongly Agree). The scores were summed for each participant. The scores range from 1-12, with higher scores indicating higher levels of PrEP Stigma.
  The higher the score, the higher the level of PrEP stigma.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow- General Health Control Arm
Number analyzed (Participants) | 69 | 63
score on a scale
  Baseline | 6.25 (2.21) | 6.78 (2.39)
  6 Weeks | 5.40 (2.55) | 6.24 (2.87)
  12 Weeks | 5.12 (2.34) | 6.0 (2.53)
Statistical Analysis 1: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 6 weeks; Test type: Superiority; p = 0.2114, Mixed Models Analysis; Slope = -0.302
Statistical Analysis 2: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 12 weeks; Test type: Superiority; p = 0.2141, Mixed Models Analysis; Slope = -0.03149

6. Secondary Outcome: Communication About PrEP
Description: Discussion of PrEP with friends, partners, or family. Communication about PrEP was measured with 2 questions, using a Likert scale ( from 1-5;1=Not at all, 5= Extremely). The scores of the 2 questions were summed for each participant.
  The scores range from 1-10, with higher the score indicating higher the level of communication about PrEP (i.e. higher scores indicates participants communicating more about PrEP).
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow- General Health Control Arm
Number analyzed (Participants) | 65 | 63
score on a scale
  Baseline | 8.42 (2.38) | 8.24 (2.29)
  6 Weeks | 9.14 (1.47) | 8.60 (1.85)
  12 Weeks | 8.94 (1.81) | 8.32 (2.14)
Statistical Analysis 1: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 6 weeks; Test type: Superiority; p = 0.0124, Mixed Models Analysis; Slope = 0.0278
Statistical Analysis 2: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 12 weeks; Test type: Superiority; p = 0.0022, Mixed Models Analysis; Slope = 0.03052

7. Secondary Outcome: PrEP Barriers
Description: Any Barriers to PrEP uptake.
  To measure barriers to PrEP uptake, 7 items were used. Each item was measured using a likert scale ( from 1-4; 1=Strongly Disagree, 4= Strongly Agree). The scores of each question were summed for each participant (scale scores ranged 1-28, with higher scores indicating higher levels of PrEP Barriers).
  The higher the score, the higher the number of PrEP Barriers.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow- General Health Control Arm
Number analyzed (Participants) | 65 | 63
score on a scale
  Baseline | 17.80 (4.28) | 18.73 (4.6)
  6 Weeks | 17.11 (5.17) | 18.76 (5.22)
  12 Weeks | 16.55 (4.92) | 17.84 (5.20)
Statistical Analysis 1: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 6 weeks; Test type: Superiority; p = 0.1021, Mixed Models Analysis; Slope = -0.05747
Statistical Analysis 2: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 12 weeks; Test type: Superiority; p = 0.133, Mixed Models Analysis; Slope = -0.05101

8. Secondary Outcome: Self-efficacy About Using PrEP
Description: Self-reported answer to questions about self-efficacy of using PrEP. There were two questions to measure self-efficacy of PrEP using a Likert scale (ranging from 1-5; 1=Not at all, 5=Extremely). The scores from both questions were summed for each participant. The scale range from 1-10 with higher scores indicating higher the levels of PrEP self-efficacy.
Time Frame: at baseline, 6 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow- General Health Control Arm
Number analyzed (Participants) | 65 | 63
score on a scale
  Baseline | 8.26 (2.39) | 8.19 (2.35)
  6 Weeks | 8.88 (1.72) | 8.49 (1.86)
  12 Weeks | 8.75 (1.97) | 8.13 (2.35)
Statistical Analysis 1: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 6 weeks; Test type: Superiority; p = 0.0818, Mixed Models Analysis; Slope = -0.0209
Statistical Analysis 2: Comparison: E-PrEP- Peer-Led Intervention About PrEP vs BxNow- General Health Control Arm; At 12 weeks; Test type: Superiority; p = 0.0334, Mixed Models Analysis; Slope = 0.03103

9. Other Pre Specified Outcome: Number of Participants With Self-reported HIV Testing
Description: Self-reported HIV testing at baseline, 6 weeks, and 12 weeks.
Time Frame: at baseline, 6 weeks, and 12 weeks
Population: Each row indicates when the participant who responded to the survey at baseline, 6 weeks, and 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow- General Health Control Arm
Number analyzed (Participants) | 81 | 71
Participants
  Baseline: 1 month | 33 | 22
  Baseline: 3 months or less | 29 | 20
  Baseline: 4 to 6 months | 10 | 16
  Baseline: 7 to 12 months | 6 | 7
  Baseline: More than 12 months | 1 | 2
  Baseline: I have never been tested for STI | 2 | 4
  6 Weeks: number analyzed (Participants) | 69 | 66
  6 Weeks: 1 month | 24 | 20
  6 Weeks: 3 months or less | 26 | 23
  6 Weeks: 4 to 6 months | 11 | 13
  6 Weeks: 7 to 12 months | 1 | 6
  6 Weeks: More than 12 months | 5 | 3
  6 Weeks: I have never been tested for STI | 2 | 1
  12 Weeks: number analyzed (Participants) | 71 | 65
  12 Weeks: 1 month | 26 | 18
  12 Weeks: 3 months or less | 31 | 19
  12 Weeks: 4 to 6 months | 9 | 15
  12 Weeks: 7 to 12 months | 0 | 7
  12 Weeks: More than 12 months | 4 | 3
  12 Weeks: I have never been tested for STI | 1 | 3

10. Other Pre Specified Outcome: Number of Participants With Self-reported Linkage-to-Care
Description: Self-reported information about health care access (i.e. going to a medical appointment).
Time Frame: at baseline, 6 weeks, and 12 weeks
Population: Each row has the number of participants who access healthcare at each time point in the "yes" category, and the number of people who did not access healthcare in the "no" category. (Baseline vs. 6 weeks vs. 12 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow- General Health Control Arm
Number analyzed (Participants) | 81 | 71
Participants
  Baseline- Visit in the past 12 months: Yes | 61 | 64
  Baseline- Visit in the past 12 months: No | 20 | 7
  6 Weeks- Visit in the past 6 weeks: number analyzed (Participants) | 69 | 66
  6 Weeks- Visit in the past 6 weeks: Yes | 40 | 41
  6 Weeks- Visit in the past 6 weeks: No | 29 | 25
  12 Weeks- Visit in the past 12 weeks: number analyzed (Participants) | 71 | 65
  12 Weeks- Visit in the past 12 weeks: Yes | 45 | 33
  12 Weeks- Visit in the past 12 weeks: No | 26 | 32

11. Other Pre Specified Outcome: Trust in the Peer by Participant
Description: The scale measure the level of trust the Participant had on the Peer's online post.
  Trust in the Peer Leader was measured using 4 questions, each scored from 1-7 (1=Strongly Disagree, 7=Strongly Agree). The score for the 4 questions was summed for each participant. The score ranged from 1-28 with higher scores indicating a higher level of trust the participant had in their Peer Leader.
Time Frame: at baseline and 6 weeks
Population: The total number of participants who completed baseline study was 81 for e-prep and 71 for control. The analysis for 6 weeks included only the people who completed the survey at each that time period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow- General Health Control Arm
Number analyzed (Participants) | 81 | 71
score on a scale
  Baseline | 16.4 (4.15) | 14.32 (4.27)
  6 Weeks: number analyzed (Participants) | 69 | 66
  6 Weeks | 16.06 (4.48) | 15.71 (4.28)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked for a period of 12 weeks.
Description: There was no risk for serious or adverse events. All of the the risk were minimal. None of the participants were at risk of mortality.
Arm/Group | E-PrEP- Peer-Led Intervention About PrEP | BxNow - General Health Campaign
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/71
Other Adverse Events (participants affected / at risk) | 0/81 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT03213366/Prot_SAP_000.pdf